CLINICAL TRIAL: NCT02488473
Title: Does Perineural Dexmedetomidine Prolong the Duration of an Adductor Canal Block When Controlling for a Systemic Effect? - A Randomised Paired Trial in Healthy Volunteers.
Brief Title: Does Perineural Dexmedetomidine Prolong Duration of a Nerve Block?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Hessel Andersen, Anesthesiologist, Staff Specialist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-JH-14; 2014-005651-89 (EudraCT Number)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Dexmedetomidine; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine + Dexmedetomidine (Experimental): Adductor Canal Block 20 ml Ropivacaine 5mg/ml + 1 ml Dexmedetomidine 100ug/ml
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine
- Ropivacaine + Placebo (Placebo Comparator): Adductor Canal Block 20 ml Ropivacaine 5mg/ml + 1 ml Saline
  Interventions: Drug: Ropivacaine; Drug: Isotonic Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 100 ug dexmedetomidine added to the ropivacaine nerveblock
  Other Names: Dexdor
  Arms: Ropivacaine + Dexmedetomidine
Drug: Ropivacaine — 20 ml Ropivacaine 5mg/ml
Drug: Isotonic Saline — Placebo
  Arms: Ropivacaine + Placebo

SUMMARY:
Brief Summary: The aim of this trial is to investigate if dexmedetomidine prolongs the duration of an adductor canal block. By using healthy volunteers the investigators can perform a bilateral adductor canal block and thereby control for a systemic effect to clarify if the effect is actually peripheral or systemic. The investigators hypothesis is that dexmedetomidine as an adjunct to a local anaesthetic prolongs the duration of a peripheral nerve block by a peripheral mechanism.

DETAILED DESCRIPTION:
Background:

Efficient pain management promoting mobilization and convalescence is essential in an ideal perioperative course. Regional nerve blocks are a central element in postoperative regimes for many patients and it is therefore important that these nerve blocks are both long lasting and efficient. This trial will investigate whether it is possible to optimize the postoperative pain management when adding dexmedetomidine to the local anaesthetic ropivacaine in peripheral nerve blocks.

The prolonging effect of using dexmedetomidine as adjunct in peripheral nerve blocks have been investigated in several studies. However, it remains uncertain whether the effect is mediated by a systemic-, a peripheral- or a combined systemic/peripheral mechanism. In this trial the adjuvating effect of dexmedetomidine will be investigated using the adductor canal block. This is a nerve block that besides being efficient as pain treatment after knee surgery, is primarily sensory, and therefore augments mobilization after total knee arthroplasty.

Method:

On the trial day the volunteers will receive bilateral adductor canal blocks. In one thigh they will receive the local anaesthetic ropivacaine 20ml 5mg/ml and placebo (saline) and in the other thigh ropivacaine 20ml 5mg/ml and dexmedetomidine 100μg. The allocation is blinded to volunteer and investigator.

The duration of the nerve block will be measured by five different tests: Temperature test, Pinprick, Pain during tonic heat stimulation, Warmth detection threshold and pain detection threshold. All tests are validated within pain research.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class 1
* Body Mass Index 18-30

Exclusion Criteria:

* Allergy to study medication
* Earlier trauma or surgery to lower limb
* Diabetes Mellitus
* Alcohol or drug abuse
* Daily intake of opioids or steroids last 4 weeks
* Daily intake of any analgesics last 48 hours Heart block Sick sinus node.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference in duration of sensory block between dexmedetomidine and placebo assessed as cold sensation with an alcohol swab | 0-36 hours
  Duration is defined as time from block performance until recovery of cold sensation to an alcohol swab, assessed every hour post-block (and every half hour when pain scores during the tonic heat stimulation test is above 0) Time for sleep will be provided.

SECONDARY OUTCOMES:
Difference between dexmedetomidine and placebo in the duration of a sensory block assessed by pin-prick | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block Time for sleep will be provided.
Difference between dexmedetomidine and placebo in the duration of a sensory block assessed as maximum pain during a tonic heat stimulation test | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block.Time for sleep will be provided. Recovery of normal sensation is defined as VAS pain scores ± 10 mm of the pre-block value. A Linear 100mm visual analogue scale (VAS) will be used.
Difference between dexmedetomidine and placebo in the duration of a sensory block assessed as warmth detection threshold | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block Time for sleep will be provided. Recovery of normal sensation is defined as detection thresholds of ± 2 degrees C of the pre-block value. Time for sleep will be provided
Difference between dexmedetomidine and placebo in the duration of a sensory block assessed as heat pain detection threshold | 0-36 hours
  Duration is defined as time from block performance until recovery of normal sensation, assessed on the hour post block. Time for sleep will be provided. Recovery of normal sensation is defined as detection thresholds of ± 2 degrees C of the pre-block value.
Difference in maximum pain scores between dexmedetomidine and placebo during block and after recovery of normal sensation. | 0-36 hours
  Pain scores during a tonic heat stimulation will be compared every hour post block and 1 h after pain scores have returned to the pre-block values. Time for sleep will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob H Andersen, MD, Principal Investigator — Department of Anesthesiology Koege Hospital
Locations (1):
- Department of Anesthesiology Koege Hospital, Koege, Denmark